CLINICAL TRIAL: NCT01381120
Title: Therapeutic Merit of Solifenacin in the Mitigation of Ureteral Stent-induced Pain and Lower Urinary Tract Symptoms (LUTS) Post Ureteroscopy for Stone Management
Brief Title: Therapeutic Merit of Solifenacin in the Mitigation of Ureteral Stent-induced Pain and Lower Urinary Tract Symptoms
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Barrie Urology Associates (Other)
Collaborators: Astellas Pharma Canada, Inc. (Industry)
Responsible Party: Principal Investigator, Dr. Joseph Zadra, Chief of Urology, RVH, Barrie Urology Associates
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARC-2010-03
Record Dates: First submitted 2010-09-02; First posted 2011-06-27 (Estimated); Results first posted 2012-08-22 (Estimated); Last update posted 2012-08-30 (Estimated); Status verified 2012-08

CONDITIONS: Flank Pain; Urinary Bladder, Overactive
Keywords: Flank Pain; Lower Urinary Tract Symptoms; LUTS; Urgency; Nocturia; Frequency; Ureteroscopy; Kidney Stones; Stent; Incontinence; VESIcare; Ureter; Urinary Bladder, Overactive; OAB; Overactive Bladder Syndrome
MeSH Terms: conditions — Flank Pain; Urinary Bladder, Overactive; Lower Urinary Tract Symptoms; Nocturia; Kidney Calculi | interventions — Solifenacin Succinate; Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VESIcare + Narcotic Painkiller (Experimental): VESIcare: Dosage form: tablet, film coated Dosage: 5 mg Frequency: daily Duration: three months Oxycodone and acetaminophen combination treatment: Dosage form: tablet, film coated Dosage: 10 mg Frequency: every 6 hours Duration: 5 - 8 days (stent inserted)
  Interventions: Drug: Solifenacin succinate treatment; Drug: Oxycodone and acetaminophen combination treatment
- Narcotic Painkiller (Active Comparator): Oxycodone and acetaminophen combination treatment: Dosage form: tablet, film coated Dosage: 10 mg Frequency: every 6 hours Duration: 5 - 8 days (stent inserted)
  Interventions: Drug: Oxycodone and acetaminophen combination treatment

INTERVENTIONS:
Drug: Solifenacin succinate treatment — Dosage form: tablet, film coated Dosage: 5 mg Frequency: daily Duration: three months
  Other Names: VESIcare
  Arms: VESIcare + Narcotic Painkiller
Drug: Oxycodone and acetaminophen combination treatment — Dosage form: tablet, film coated Dosage: 10 mg Frequency: every 6 hours Duration: 5 - 8 days (stent inserted)

SUMMARY:
Most ureteral stent insertions follow ureteroscopy procedures for stone management. Stents are essentially designed to prevent the blockage of the ureter. Such blockage is often a result of inflammation caused by ureteroscopy procedures. The stent provides a secure passageway for urine as it travels from the kidneys to the bladder, circumventing potential urinary retention. In our community, only one kind of stent is used, and it is manufactured by Bard. Standard protocol involves the removal of the stent 5 to 8 days following insertion. If stenting is required for greater than 8 days, special accommodations will be made for you in this study.

Unfortunately, pain and lower urinary tract symptoms are often associated with the insertion and removal of stents. It is our goal to determine whether VESIcare is capable of relieving such symptoms.

As a prospective member of this study, you will be asked to complete three surveys. The first survey will ask you about your experiences of urinary urgency and pain before your surgery. If you are an emergency patient, you will be asked to remember your condition before the surgery, completing this questionnaire at your first post-op visit. If you are not an emergency patient, this survey will be completed before your surgery. If your stent is removed within 5 to 8 days of surgery, you will be asked to complete the second survey at the time of removal. You will then complete the final survey at a scheduled post-operative check-up 4 to 5 weeks later. If your stent remains inserted for greater than 8 days after surgery, you will be asked to complete the second survey 3 to 4 days after your stent was inserted. You will then complete the final survey, 7 to 8 weeks post-op.

Throughout this study, both VESIcare and non-VESIcare patients will be important in determining whether VESIcare truly is capable of relieving stent pain. As such, you will be randomly assigned to one of the two groups, those receiving VESIcare, and those who are not.

ELIGIBILITY:
Subject inclusion criteria.

1. Post-ureteroscopy for stone management.
2. Stent inserted for more than 5 days.
3. No significant flank pain or LUTS prior to kidney stones/stent insertion.
4. Complete agreement with and signing of Informed Consent form.

Subject exclusion criteria.

1. Significant flank pain or LUTS prior to kidney stones/stent insertion.
2. Currently taking antimuscarinics or α1 blockers.
3. Patients with urinary retention, dependent on dialysis, gastroparesis or narrow angle glaucoma.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2010-10; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Zadra, MD CM FRCSC, Principal Investigator — Barrie Urology Associates - The Male/Female Health and Research Centre
Locations (1):
- Barrie Urology Associates - The Male/Female Health and Research Centre, Barrie, Ontario, Canada

REFERENCES:
- [Background] Mendez-Probst CE, Fernandez A, Denstedt JD. Current status of ureteral stent technologies: comfort and antimicrobial resistance. Curr Urol Rep. 2010 Mar;11(2):67-73. doi: 10.1007/s11934-010-0091-y. PMID 20425092
- [Background] Wang CJ, Huang SW, Chang CH. Effects of specific alpha-1A/1D blocker on lower urinary tract symptoms due to double-J stent: a prospectively randomized study. Urol Res. 2009 Jun;37(3):147-52. doi: 10.1007/s00240-009-0182-8. Epub 2009 Mar 10. PMID 19277623
- [Background] Damiano R, Autorino R, De Sio M, Giacobbe A, Palumbo IM, D'Armiento M. Effect of tamsulosin in preventing ureteral stent-related morbidity: a prospective study. J Endourol. 2008 Apr;22(4):651-6. doi: 10.1089/end.2007.0257. PMID 18338955
- [Background] Park SC, Jung SW, Lee JW, Rim JS. The effects of tolterodine extended release and alfuzosin for the treatment of double-j stent-related symptoms. J Endourol. 2009 Nov;23(11):1913-7. doi: 10.1089/end.2009.0173. PMID 19814699
- [Background] Joshi HB, Newns N, Stainthorpe A, MacDonagh RP, Keeley FX Jr, Timoney AG. Ureteral stent symptom questionnaire: development and validation of a multidimensional quality of life measure. J Urol. 2003 Mar;169(3):1060-4. doi: 10.1097/01.ju.0000049198.53424.1d. PMID 12576846

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | VESIcare + Narcotic Painkiller | Narcotic Painkiller
Started | 50 | 27
Completed | 39 | 18
Not Completed | 11 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VESIcare + Narcotic Painkiller | Narcotic Painkiller | Total
Number analyzed (Participants) | 50 | 27 | 77
Age Continuous [Mean (Standard Deviation); unit: years] | 50.81 (12.36) | 57.54 (18.73) | 53 (15.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 13 | 46
  Male | 17 | 14 | 31

OUTCOME MEASURES:

1. Primary Outcome: Change in Post-ureteroscopy Stent-induced Pain
Description: Measured through the use of the ureteral stent symptom questionnaire. Patients reported pain on a scale of 0 to 10 (0 being the absence of pain and 10 being the most excruciating pain of their life). The questionnaire was administered a couple days post-op and once again several weeks later. The mean difference (baseline minus 3 months) on this continuous scale was used for this outcome measure.
Time Frame: Baseline and 3 months.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | VESIcare + Narcotic Painkiller | Narcotic Painkiller
Number analyzed (Participants) | 39 | 18
units on a scale | 4.61 [3.75 to 5.46] | 3.11 [1.63 to 4.60]

2. Secondary Outcome: Change in Post-ureteroscopy Stent-induced Lower Urinary Tract Symptoms.
Description: Measured through the use of the ureteral stent symptom questionnaire. Patients reported symptoms on a scale of 1 to 5 (1 being the absence of symptoms and 5 being very debilitating symptoms). The questionnaire was administered a couple days post-op and once again several weeks later. The mean difference (baseline minus 3 months) on this continuous scale was used for this outcome measure.
Time Frame: Baseline and three months.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | VESIcare + Narcotic Painkiller | Narcotic Painkiller
Number analyzed (Participants) | 39 | 18
units on a scale | 1.90 [1.60 to 2.21] | 1.13 [0.82 to 1.43]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for the duration of the study (October 2010 - June 2012)
Description: Non-serious events were not recorded. Patients were encouraged to contact the study coordinator if they experienced any serious adverse events.
Arm/Group | VESIcare + Narcotic Painkiller | Narcotic Painkiller
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/27
Other Adverse Events (participants affected / at risk) | 0/50 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No